CLINICAL TRIAL: NCT01965405
Title: Behavioral Smoking Cessation Treatment for People Living With HIV/AIDS
Brief Title: Smoking Cessation for People Living With HIV/AIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Ledgerwood, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA034537-01A1 (NIH); 1R01DA034537-01A1 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-18 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: HIV; AIDS; Nicotine Dependence
Keywords: HIV; AIDS; Nicotine Dependence; Smoking; Smoking cessation; Contingency Management
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1: Standard of Care (A) (Experimental): Brief counseling and bupropion
  Interventions: Drug: Bupropion; Behavioral: Brief Counseling
- Phase 1: Standard of Care (B) (Experimental): Brief counseling, bupropion, and brief high-magnitude prize contingency management.
  Interventions: Drug: Bupropion; Behavioral: Brief Counseling; Behavioral: High-magnitude prize contingency management
- Phase 2a Non-Responders (A) (Experimental): Bupropion, continued counseling, monitored support to quit smoking.
  Interventions: Drug: Bupropion; Behavioral: Brief Counseling; Behavioral: Monitored support to quit smoking
- Phase 2a: Non-Responders (B) (Experimental): Bupropion, monitored support to quit smoking, prize contingency management for abstinence.
  Interventions: Drug: Bupropion; Behavioral: Monitored support to quit smoking; Behavioral: Prize contingency management for abstinence
- Phase 2b: Responders (A) (Experimental): Bupropion, no additional treatment.
  Interventions: Drug: Bupropion; Behavioral: No additional treatment
- Phase 2b: Responders (B) (Experimental): Bupropion, continued monitoring and low intensity prize contingency management.
  Interventions: Drug: Bupropion; Behavioral: Monitored support to quit smoking; Behavioral: Low intensity prize contingency management

INTERVENTIONS:
Drug: Bupropion — Participant will receive a prescription for Bupropion hydrochloride and will self-administer according to dosage instructions from the study psychiatrist.
  Other Names: Bupropion hydrochloride; Wellbutrin; Zyban
Behavioral: Brief Counseling — Participants are provided with brief counseling for smoking cessation.
  Arms: Phase 1: Standard of Care (A); Phase 1: Standard of Care (B); Phase 2a Non-Responders (A)
Behavioral: High-magnitude prize contingency management — Prize based contingency management condition in which participants have the chance to win incentives (prizes) when they provide biological test results (expired carbon monoxide and cotinine) that are negative for recent smoking.
  Arms: Phase 1: Standard of Care (B)
Behavioral: Monitored support to quit smoking — Brief supportive sessions and monitoring of smoking cessation efforts.
  Arms: Phase 2a Non-Responders (A); Phase 2a: Non-Responders (B); Phase 2b: Responders (B)
Behavioral: No additional treatment — No additional treatment will be given.
  Arms: Phase 2b: Responders (A)
Behavioral: Prize contingency management for abstinence — Prize based contingency management condition in which participants have the chance to win incentives (prizes) when they provide biological test results (expired carbon monoxide and cotinine) that are negative for recent smoking.
  Arms: Phase 2a: Non-Responders (B)
Behavioral: Low intensity prize contingency management — Prize based contingency management condition in which participants have the chance to win incentives (prizes) when they provide biological test results (expired carbon monoxide and cotinine) that are negative for recent smoking.
  Arms: Phase 2b: Responders (B)

SUMMARY:
In this proposed study with People Living with HIV/AIDS (PLWHA), we will use a stepped care model called a Sequential Multiple Assignment Randomized Trial (SMART) to examine the efficacy of low- and high-intensity smoking cessation treatments for nicotine dependent PLWHA that incorporate the current standard of care and prize-based contingency management. Intervention will be administered in a community-based HIV integrated care clinic in downtown Detroit, which has the highest prevalence rates of HIV/AIDS and smoking in Michigan. Phase 1 will last 4 weeks, and will involve brief intervention to help participants stop smoking. For phase 2, participants will be assigned to different study arms depending on whether they are Responders (reduced their smoking) or Non-responders (continued to smoke).

1. Phase 1: We hypothesize that brief high-magnitude prize contingency management will result in greater reduction in smoking than standard of care alone.
2. Phase 2a: We hypothesize that non-responders who are assigned to contingency management will be more likely to reduce their smoking throughout treatment and to abstain from smoking at all follow-up points.
3. Phase 2b: We hypothesize that responders who are assigned to monitoring and low-magnitude prize contingency management will be more likely to maintain their reduced or abstinent smoking status at all follow-up time-points.

DETAILED DESCRIPTION:
All research related activities will take place at the Tolan Park Medical Building located at 3901 Chrysler Service Dr, Detroit, 48201.

Participants in Phase 1 will be randomized to one of two brief interventions based on standard of care guidelines (SoC): A) brief counseling and bupropion (SoC); or B) SoC plus brief high-magnitude prize CM (HM-CM). At the end of Phase 1, participants will be classified as responders or non-responders on the basis of smoking reduction/abstinence. All participants will continue to receive bupropion. Non-responders will enter Phase 2a and be randomly assigned to: A) continued counseling and monitoring support to quit smoking (MS); or B) MS plus prize CM for abstinence (MS+CM). Phase 1 responders will be entered into Phase 2b and randomly assigned to: A) no additional treatment (NAT); or B) Continued monitoring and low intensity prize CM (LI-CM). The primary dependent variables will include cotinine and carbon monoxide (CO) levels, and longest duration of abstinence from cigarettes. Seven-day point prevalence will be used to assess outcome at post-treatment, 6-month and 12-month follow-up points.

Participants will be paid $35 for intake and $25 for each follow-up interview, which will occur at post-phase 1, post-phase 2, and 6-months and 12-months after treatment initiation. Some assessments as well as treatment sessions will be recorded to ensure data quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to read and understand English
3. Smoke more than 10 cigarettes/day
4. Patient enrolled in the HIV clinic with HIV or AIDS diagnosis

Exclusion Criteria:

1. Are actively suicidal or have uncontrolled manic or psychotic symptoms requiring immediate care
2. Are in recovery for pathological gambling (PG)
3. Have contraindications for bupropion treatment (e.g., presence of epilepsy or other seizure disorder, use of monoamine oxidase inhibitors or other antidepressants, presence of eating disorders or very low weight)
4. Are already participating in other smoking cessation interventions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Urinary Cotinine | Change from baseline: weekly in treatment phase 1; between 0 to 16 times during treatment phase 2 (non-responders meet 16 times; responders meet 0 or 6 times depending on group); Follow-up interviews (Post-phase 1, Post-phase 2, 6-months and 12-months)
  Urinary cotinine is a metabolite of nicotine, and can be detected in urine. The presence of cotinine in urine shows recent cigarette smoking. Cotinine is measured using an instant test that give a score from 0 to 6 on a semi-quantitative scale. Declining scores show an individual has stopped or significantly reduced their smoking.
Longest Duration of Continuous Abstinence | Change from baseline: Weekly through treatment phase 1; between 0 to 16 times during treatment phase 2 (non-responders meet 16 times; responders meet 0 or 6 times depending on group)
  This is the longest period of consecutive days during treatment where the participant has not smoked. Longest duration of abstinence is calculated through self-report of smoking abstinence verified by scores on biological measures (negative scores on carbon monoxide or urinary cotinine tests).
Seven-Day Point-Prevalence | Follow-up interviews: Post-phase 1, Post-phase 2, 6-months and 12-months after treatment initiation.
  At each follow-up assessment, participants will be asked if they had smoked in the preceding seven days. They will also participate in cotinine and carbon monoxide testing. Negative scores are given when the participant reports no smoking and all tests are negative.
Carbon Monoxide Results | Change from baseline: weekly in treatment phase 1; between 0 to 16 times during treatment phase 2 (non-responders meet 16 times; responders meet 0 or 6 times depending on group); Follow-up interviews (Post-phase 1, Post-phase 2, 6-months and 12-months)
  Participants will provide breath carbon monoxide samples at each visit by blowing into a hand-held carbon monoxide reader. Carbon monoxide is produced when substances (such as cigarettes) are burned. Thus this test can show if an individual has been smoking recently.

CONTACTS AND LOCATIONS:
Overall Officials: David Ledgerwood, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

REFERENCES:
- [Derived] Ledgerwood DM, Lundahl LH, Greenwald MK, Cohn J, Arfken CL. Prize-Based Incentives for Smoking Cessation Among People With HIV: A Sequential Multiple Assignment Randomized Trial. Nicotine Tob Res. 2025 Apr 22;27(5):893-902. doi: 10.1093/ntr/ntae243. PMID 39404754